CLINICAL TRIAL: NCT01796301
Title: An Open-label, Randomized, Teriparatide-controlled Study to Evaluate the Effect of Treatment With Romosozumab in Postmenopausal Women With Osteoporosis Previously Treated With Bisphosphonate Therapy
Brief Title: An Open-label Study to Evaluate the Effect of Treatment With Romosozumab or Teriparatide in Postmenopausal Women
Acronym: STRUCTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080289; 2012-002948-24 (EudraCT Number)
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — romosozumab; Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Romosozumab (Experimental): Participants received 210 mg romosozumab administered by subcutaneous injection once a month for 12 months.
  Interventions: Drug: Romozosumab
- Teriparatide (Active Comparator): Participants received 20 μg/day teriparatide administered by subcutaneous injection for 12 months.
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Romozosumab — Administered by subcutaneous injection once a month.
  Other Names: AMG 785
  Arms: Romosozumab
Drug: Teriparatide — Administered by subcutaneous injection once a day.
  Other Names: Forteo; Forsteo
  Arms: Teriparatide

SUMMARY:
The primary objective of the study was to evaluate the effect of 12 months of treatment with romosozumab compared with teriparatide on total hip bone mineral density (BMD) in postmenopausal women with osteoporosis who were previously treated with bisphosphonate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, aged ≥ 55 to ≤ 90.
* Received oral bisphosphonate therapy for at least 3 years immediately prior to screening
* BMD T-score ≤ -2.50 at the lumbar spine, total hip or femoral neck
* History of nonvertebral fracture after age 50, or vertebral fracture.

Exclusion Criteria:

* Use of other agents affecting bone metabolism including Strontium ranelate, fluoride (for osteoporosis), odanacatib (MK-0822) or any other cathepsin K inhibitor, IV bisphosphonates, denosumab, teriparatide (TPTD) or any parathyroid hormone (PTH) analogs, Systemic oral or transdermal estrogen, selective estrogen receptor modulators (SERMs), activated vitamin D3, vitamin K2, calcitonin, tibolone, cinacalcet, systemic glucocorticosteroids:
* History of metabolic or bone disease (except osteoporosis) that may interfere with the interpretation of study results, such as sclerosteosis, Paget's disease, rheumatoid arthritis, osteomalacia, osteogenesis imperfecta, osteopetrosis, ankylosing spondylitis, Cushing's disease, hyperprolactinemia, and malabsorption syndrome.
* Vitamin D insufficiency, defined as 25 (OH) vitamin D levels < 20 ng/mL, as determined by the central laboratory.
* Current hyper- or hypocalcemia
* Current, uncontrolled hyper- or hypothyroidism

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (44):
- United States (4):
  - Research Site, Gainesville, Georgia
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
- Argentina (2):
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
- Belgium (4):
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
- Colombia (2):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
- Czechia (5):
  - Research Site, Brno
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Praha 11 - Chodov
  - Research Site, Uherské Hradiště
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Aarhus C
  - Research Site, Ballerup Municipality
  - Research Site, Esbjerg
  - Research Site, Hillerød
  - Research Site, Hvidovre
  - Research Site, Odense
- Research Site, Budapest, Hungary
- Poland (4):
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Spain (5):
  - Research Site, Granada, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, LHospitalet de Llobregat, Catalonia
  - Research Site, Pozuelo de Alarcón, Madrid
  - Research Site, Madrid
- United Kingdom (6):
  - Research Site, Cardiff
  - Research Site, Chorley
  - Research Site, Liverpool
  - Research Site, Northwood
  - Research Site, Reading
  - Research Site, Sidcup

REFERENCES:
- [Background] Langdahl BL, Libanati C, Crittenden DB, Bolognese MA, Brown JP, Daizadeh NS, Dokoupilova E, Engelke K, Finkelstein JS, Genant HK, Goemaere S, Hyldstrup L, Jodar-Gimeno E, Keaveny TM, Kendler D, Lakatos P, Maddox J, Malouf J, Massari FE, Molina JF, Ulla MR, Grauer A. Romosozumab (sclerostin monoclonal antibody) versus teriparatide in postmenopausal women with osteoporosis transitioning from oral bisphosphonate therapy: a randomised, open-label, phase 3 trial. Lancet. 2017 Sep 30;390(10102):1585-1594. doi: 10.1016/S0140-6736(17)31613-6. Epub 2017 Jul 26. PMID 28755782
- [Background] Takada J, Dinavahi R, Miyauchi A, Hamaya E, Hirama T, Libanati C, Nakamura Y, Milmont CE, Grauer A. Relationship between P1NP, a biochemical marker of bone turnover, and bone mineral density in patients transitioned from alendronate to romosozumab or teriparatide: a post hoc analysis of the STRUCTURE trial. J Bone Miner Metab. 2020 May;38(3):310-315. doi: 10.1007/s00774-019-01057-1. Epub 2019 Nov 9. PMID 31707465
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 46 sites in North America, Latin America, and Europe. Participants were enrolled from 31 January 2013 to 29 April 2014.
Pre-assignment Details: A total of 777 subjects were screened for participation; 341 (43.9%) were excluded prior to randomization, primarily due to not meeting inclusion/exclusion criteria (306 [39.4%] subjects). A total of 436 participants were randomized into the study.
Period: Overall Study
Arm/Group | Teriparatide | Romosozumab
Started | 218 | 218
Received Treatment | 214 | 218
Completed | 200 | 198
Not Completed | 18 | 20
Not completed — Withdrawal by Subject | 15 | 15
Not completed — Lost to Follow-up | 3 | 3
Not completed — Death | 0 | 1
Not completed — Decision by Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Romosozumab | Total
Number analyzed (Participants) | 218 | 218 | 436
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (7.7) | 71.8 (7.4) | 71.5 (7.5)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 48 | 50 | 98
  ≥ 65 to < 75 years | 96 | 83 | 179
  ≥ 75 years | 74 | 85 | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 218 | 436
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 196 | 191 | 387
  Other | 18 | 23 | 41
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 2 | 0 | 2
  Multiple | 1 | 0 | 1
Prior Fracture [Count of Participants; unit: Participants]
  Yes | 217 | 218 | 435
  No | 1 | 0 | 1
Lumbar Spine BMD T-score [Mean (Standard Deviation); unit: T-score] — The T-score is the bone mineral density (BMD) at the site when compared to that of a healthy thirty-year-old. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score | -2.87 (1.04) | -2.83 (1.10) | -2.85 (1.07)
Total Hip BMD T-score [Mean (Standard Deviation); unit: T-score] | -2.21 (0.72) | -2.27 (0.75) | -2.24 (0.74)
Femoral Neck BMD T-score [Mean (Standard Deviation); unit: T-score] | -2.43 (0.66) | -2.49 (0.67) | -2.46 (0.66)
Serum Type 1 Collagen C-telopeptide (sCTX) [Mean (Standard Deviation); unit: ng/L] | 260.1 (124.9) | 252.3 (136.4) | 256.2 (130.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline Through Month 12 in Total Hip Bone Mineral Density (BMD)
Description: Bone mineral density was measured by dual-energy X-ray absorptiometry (DXA). Percent change from baseline through month 12 is the average of the treatment effect at months 6 and 12.
Time Frame: Baseline, month 6 and month 12
Population: The primary efficacy analysis set includes randomized participants with a non-missing baseline and at least one post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 209 | 206
percent change | -0.6 (0.2) | 2.6 (0.2)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; The primary analysis to assess the treatment difference (Romosozumab - Teriparatide) employed a linear mixed effects model for repeated measures. The model included main effects for treatment group, visit (categorical), baseline sCTX, baseline hip DXA BMD value, machine type (categorical), and machine type-by-baseline value interaction (to adjust for the effect of machine type on baseline DXA BMD value) as fixed main effects using an unstructured within-subject variance-covariance structure; Test type: Superiority — A two-step, step-down, fixed-sequential testing procedure was used to test the primary and key secondary efficacy endpoints for the comparison of romosozumab to teriparatide in the order presented for multiplicity adjustment to maintain the overall significance level at 0.05. The Key Secondary Efficacy Endpoints are the first 8 secondary endpoints reported below; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.2, 95% CI 2-sided [2.7 to 3.8], Standard Error of Mean 0.3

2. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 6
Description: Bone mineral density was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and month 6
Population: The primary efficacy analysis set with values at baseline and month 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 203 | 203
percent change | -0.8 (0.2) | 2.3 (0.2)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; Treatment difference (Romosozumab - Teriparatide) was analyzed using a linear mixed effects model for repeated measures adjusting for treatment, visit, baseline serum type 1 collagen C-telopeptide value, baseline BMD value, machine type, baseline BMD value-by machine type interaction, treatment-by-visit interaction, and using an unstructured variance covariance structure; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.1, 95% CI 2-sided [2.5 to 3.7], Standard Error of Mean 0.3

3. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 12
Description: Bone mineral density was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and month 12
Population: The primary efficacy analysis set with values at baseline and month 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 202 | 197
percent change | -0.5 (0.2) | 2.9 (0.2)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.4, 95% CI 2-sided [2.8 to 4.0], Standard Error of Mean 0.3

4. Secondary Outcome: Percent Change From Baseline in Cortical BMD by Quantitative Computed Tomography (QCT) at the Total Hip at Month 6
Description: Cortical BMD was measured by quantitative computed tomography (QCT) at the total hip.
Time Frame: Baseline and month 6
Population: The primary efficacy analysis set with values at baseline and month 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 156 | 163
percent change | -2.7 (0.2) | 0.7 (0.2)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; Treatment difference (Romosozumab - Teriparatide) was analyzed using a linear mixed effects model for repeated measures adjusting for treatment, visit, baseline serum type 1 collagen C-telopeptide value, parameter baseline value, treatment-by visit interaction, and using an unstructured variance covariance structure; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.4, 95% CI 2-sided [2.8 to 4.0], Standard Error of Mean 0.3

5. Secondary Outcome: Percent Change From Baseline in Cortical BMD by QCT at the Total Hip at Month 12
Description: Cortical BMD was measured by quantitative computed tomography (QCT) at the total hip.
Time Frame: Baseline and month 12
Population: The primary efficacy analysis set with values at baseline and month 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 159 | 163
percent change | -3.6 (0.3) | 1.1 (0.3)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 4.6, 95% CI 2-sided [3.9 to 5.3], Standard Error of Mean 0.4

6. Secondary Outcome: Percent Change From Baseline in Integral BMD by QCT at the Total Hip at Month 6
Description: Integral BMD was measured by quantitative computed tomography (QCT) at the total hip.
Time Frame: Baseline and month 6
Population: The primary efficacy analysis set with values at baseline and month 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 156 | 163
percent change | -0.8 (0.2) | 2.3 (0.2)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.1, 95% CI 2-sided [2.5 to 3.6], Standard Error of Mean 0.3

7. Secondary Outcome: Percent Change From Baseline in Integral BMD by QCT at the Total Hip at Month 12
Description: Integral BMD was measured by quantitative computed tomography (QCT) at the total hip.
Time Frame: Baseline and month 12
Population: The primary efficacy analysis set with values at baseline and month 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 159 | 163
percent change | -0.2 (0.2) | 3.4 (0.2)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.6, 95% CI 2-sided [2.9 to 4.2], Standard Error of Mean 0.3

8. Secondary Outcome: Percent Change From Baseline in Estimated Strength at the Total Hip at Month 6
Description: Total hip estimated strength was assessed by finite element analysis (FEA) of QCT scans.
Time Frame: Baseline and month 6
Population: The primary efficacy analysis set with values at baseline and month 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 163 | 164
percent change | -1.0 (0.2) | 2.1 (0.2)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.1, 95% CI 2-sided [2.4 to 3.8], Standard Error of Mean 0.3

9. Secondary Outcome: Percent Change From Baseline in Estimated Strength at the Total Hip at Month 12
Description: Total hip estimated strength was assessed by finite element analysis (FEA) of QCT scans.
Time Frame: Baseline and month 12
Population: The primary efficacy analysis set with values at baseline and month 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 155 | 159
percent change | -0.7 (0.4) | 2.5 (0.4)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.2, 95% CI 2-sided [2.1 to 4.3], Standard Error of Mean 0.6

10. Secondary Outcome: Percent Change From Baseline in Total Hip Integral Bone Mineral Content (BMC) by QCT at Month 6
Description: Total hip integral BMC was measured using quantitative computed tomography (QCT).
Time Frame: Baseline and month 6
Population: The primary efficacy analysis set with values at baseline and month 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 156 | 163
percent change | -0.7 (0.2) | 2.4 (0.2)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.1, 95% CI 2-sided [2.6 to 3.6], Standard Error of Mean 0.3

11. Secondary Outcome: Percent Change From Baseline in Total Hip Integral Bone Mineral Content (BMC) by QCT at Month 12
Description: Total hip integral BMC was measured using quantitative computed tomography (QCT).
Time Frame: Baseline and month 12
Population: The primary efficacy analysis set with values at baseline and month 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 159 | 163
percent change | 0.0 (0.2) | 3.6 (0.2)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.6, 95% CI 2-sided [2.9 to 4.2], Standard Error of Mean 0.3

12. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Month 6
Description: Bone mineral density was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and month 6
Population: The primary efficacy analysis set with values at baseline and month 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 203 | 203
percent change | -1.1 (0.3) | 2.1 (0.3)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.2, 95% CI 2-sided [2.5 to 3.9], Standard Error of Mean 0.4

13. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Month 12
Description: Bone mineral density was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and month 12
Population: The primary efficacy analysis set with values at baseline and month 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 202 | 197
percent change | -0.2 (0.3) | 3.2 (0.3)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.4, 95% CI 2-sided [2.6 to 4.2], Standard Error of Mean 0.4

14. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 6
Description: Bone mineral density was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and month 6
Population: The primary efficacy analysis set with values at baseline and month 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 204 | 203
percent change | 3.5 (0.3) | 7.2 (0.3)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 3.8, 95% CI 2-sided [2.9 to 4.6], Standard Error of Mean 0.4

15. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 12
Description: Bone mineral density was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and month 12
Population: The primary efficacy analysis set with values at baseline and month 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Teriparatide | Romosozumab
Number analyzed (Participants) | 201 | 197
percent change | 5.4 (0.4) | 9.8 (0.4)
Statistical Analysis 1: Comparison: Teriparatide vs Romosozumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Linear mixed effects repeated measures; Treatment difference = 4.4, 95% CI 2-sided [3.4 to 5.4], Standard Error of Mean 0.5

ADVERSE EVENTS:
Time Frame: 12 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Teriparatide | Romosozumab
Serious Adverse Events (participants affected / at risk) | 23/214 | 17/218
Other Adverse Events (participants affected / at risk) | 76/214 | 79/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teriparatide (N=214) | Romosozumab (N=218)
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bifascicular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Radicular pain (Nervous system disorders) | 1 | 0
Radicular syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Medical device removal (Surgical and medical procedures) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Teriparatide (N=214) | Romosozumab (N=218)
Nasopharyngitis (Infections and infestations) | 22 | 28
Upper respiratory tract infection (Infections and infestations) | 9 | 11
Fall (Injury, poisoning and procedural complications) | 5 | 12
Hypercalcaemia (Metabolism and nutrition disorders) | 22 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 11
Headache (Nervous system disorders) | 9 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.